CLINICAL TRIAL: NCT01551277
Title: Use of Breath Stacking Technique on Regional Ventilation in Box Chest in Women With Morbid Obesity: Clinical Trial Controlled and Randominzado
Brief Title: Use of Breath Stacking Technique on Regional Ventilation in Box Chest in Women With Morbid Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Daniella Cunha Brandao, PhD, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: jaqueline 01
Record Dates: First submitted 2012-03-08; First posted 2012-03-12 (Estimated); Last update posted 2012-03-12 (Estimated); Status verified 2012-03

CONDITIONS: Morbidly Obese

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (Placebo Comparator)
  Interventions: Other: Placebo-BREATH STACKING
- BREATH STACKING (Experimental)
  Interventions: Other: BREATH STACKING

INTERVENTIONS:
Other: Placebo-BREATH STACKING — The control group used the same circuit in the intervention group, but without occlusion of the expiratory branch and followed the same protocol to capture the images, ie, basal respiration for five minutes, then three periods of breathing through the mask, the equivalent time the period of technical BS, and five minutes of respiration. The volunteers were instructed to maintain respiration during the period they were using the mask.
  Arms: Control Group
Other: BREATH STACKING — In the intervention group used a silicon mask, involving the nose and mouth with two outputs, one containing the Wright spirometer MARK 8 analog output and the other was occluded. It was explained that the mask would only allow the air entering during inspiration, and that should inspire the volunteer gradually filling the lungs with air until you feel that completely filled with an average time of 20 seconds, as shown in figure 1 obtained during the method of BS. The end of the technique would be in two situations: when the volunteer asked for it through a hand gesture, or when prearranged by Wright spirometer, was observed by the researcher that there was no change in the inspired volume.
  Arms: BREATH STACKING

SUMMARY:
Objectives: To evaluate the effects of the technique of Breath Stacking (BS) in the distribution of ventilation in the chest in women with morbid obesity. Methods: Randomized clinical trial, blinded, and controlled with 32 women (BMI ≥ 40kg/m2), separated into two groups: control (GC) with n = 16 and 41.94 ± 9.38 years and group Breath Stacking (GBS) , n = 16 and 40.38 ± 10.16 years. Optoelectronic plethysmography (POE) was used to assess lung ventilation. For the BS technique was used to mask the expiratory branch occluded and Wright spirometer. GBS held three techniques with an interval of three minutes. The GC used the same circuit without the occlusion of the expiratory branch. Results: GBS was found to be higher in the contribution of tidal volume (VT) into the chest circumference (p = 0.04) and decrease in abdominal compartment (p = 0.03), whereas the CG showed no difference in distribution. Spirometric variables: FEV1 (%), FVC (%), FEV1/FVC (%), VC and CI showed no difference before and after the technical BS and GBS in the GC. Conclusions: The technique BS altered the distribution pattern of regional ventilation, resulting in greater contribution in lung volume in the lower rib cage, corresponding to activity of the diaphragm, with redistribution of volume between compartments.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 19-60 years
* BMI ≥ 40 kg/m2

Exclusion Criteria:

* Women with chronic lung disease
* Smokers
* Neuromuscular disease
* Disability in performing the procedures

Ages: 19 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2010-03; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Chest wall regional volume | ten months
  We considered as primary outcome regional tidal volumes: total current volume of the chest cavity (Vc), changes in tidal volume of pulmonary rib cage (ΔVc, ctp), tidal volume variation of the abdominal rib cage (ΔVc, CTA) and abdominal tidal volume (ΔVc, ab), and secondary outcome Inspiratory capacity (IC).

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de Pernambuco, Recife, Pernambuco, Brazil

REFERENCES:
- [Result] Cala SJ, Kenyon CM, Ferrigno G, Carnevali P, Aliverti A, Pedotti A, Macklem PT, Rochester DF. Chest wall and lung volume estimation by optical reflectance motion analysis. J Appl Physiol (1985). 1996 Dec;81(6):2680-9. doi: 10.1152/jappl.1996.81.6.2680. PMID 9018522
- [Result] Chlif M, Keochkerian D, Choquet D, Vaidie A, Ahmaidi S. Effects of obesity on breathing pattern, ventilatory neural drive and mechanics. Respir Physiol Neurobiol. 2009 Sep 30;168(3):198-202. doi: 10.1016/j.resp.2009.06.012. Epub 2009 Jun 24. PMID 19559105